CLINICAL TRIAL: NCT02452411
Title: Differential Efficacy of Two Ways of Applying Homework Assignments in the Treatment of Adjustment Disorders: Application Supported by Information and Communication Technologies Versus Traditional Application
Brief Title: Efficacy of Two Ways of Applying Homework Assignments in the Treatment of Adjustment Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UJaumeI010
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Adjustment Disorders
Keywords: Internet; Adjustment disorders; Homework assignments; Cognitive-Behavioral treatment; Online therapy; Emotional Regulation; ICT's
MeSH Terms: conditions — Adjustment Disorders; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homework assignments using TEO system (Experimental): Experimental: Homework assignments using TEO system. It is an internet-based system which allows the therapist to create homework sessions using multimedia materials (videos, images, texts, and narratives) and to offer and present this material to the patients through the Internet. Participants receive a CBT treatment for adjustment disorder supported by virtual reality and they do the homework assignments component using TEO at home over the Internet.
  Interventions: Behavioral: Cognitive Behavioral Treatment approach supported by virtual reality and positive psychology strategies.
- Homework assignments using Traditional method (Experimental): The traditional way of applying homework assignments consists of reading and writing materials and audio session records. Participants receive a CBT treatment supported by virtual reality for adjustment disorder and they do the homework assignments component at home using traditional materials.
  Interventions: Behavioral: Cognitive Behavioral Treatment approach supported by virtual reality and positive psychology strategies.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Treatment approach supported by virtual reality and positive psychology strategies. — The CBT program consists of 6 weekly sessions (and 2 additional ones depending on the patient's needs) with the following main therapeutic components: educational component, exposure/processing of the stressful event with VR (EMMA's World) and relapse prevention. EMMA's World is an open and flexible VR system that uses symbols (e.g., 3D-objects, pictures, sounds) to reflect and evoke the negative emotions associated to the stressful event. Also, several strategies from Positive Psychology (e.g., My best virtues or strengths exercise) and others based on Neimeyer's (2000) suggestions for pathological grief (e.g., projection letter to the future) are also included in the protocol.
  Other Names: Psychological Treatment for Adjustment Disorders

SUMMARY:
The purpose of this study is to determine the differential efficacy of two ways of applying homework assignments in the treatment of Adjustment Disorders: 1) using an Internet-based emotional regulation therapy system (TEO) and 2) in the traditional way (using reading and audio materials).

The principal hypothesis is that both treatment conditions (TEO and Traditional) will show a similar efficacy. All participants will improve significantly on all outcome measures, regardless the type of homework assigned (TEO or Traditional) with no differences between them.

DETAILED DESCRIPTION:
Adjustment Disorders (AD) are very prevalent in primary care and hospital settings. The available data indicate that the percentage of adults suffering from AD in primary care ranges from 5% to 21%. Furthermore, AD is an important public mental health problem in economic terms. Very frequently the distress and activity deterioration associated to this problem result in a decrease of work performance, causing a high percentage of sick leaves. However, nowadays there are no evidence-based psychological treatments for this problem, and only general treatment guidelines are available for this problem. For these reason, a Cognitive-Behavioral Treatment (CBT) supported by Virtual Reality (VR; EMMA system) was developed and has already shown its utility to treat this disorder. Information and Communication Technologies (ICTs) are useful tools for offer and improve therapeutic services. VR offers a safe and flexible environment in where the person can explore and manage their problems in a controlled and gradual way. Computerized programs allow reducing the contact time between therapist and patient, so it can reach patients who would not receive treatment otherwise. ICTs have been mainly used within the therapeutic context; specifically many studies have been centered on how to use the technologies to deliver the treatment. As far as the investigators know, no study analyzes the ICTs contribution in the homework assignments field. CBT approach provides a crucial role to homework assignments because it allows reinforcing and supporting the patients along the therapy. More studies examining the utility of the application of ICTs for the treatment of AD are needed. Furthermore, the application of the homework assignments component through the Internet is also relevant. It is necessary an adaptive and flexible system that allows adjusting the therapeutic homework on every patient's characteristics and needs, attending to the specific meaning of his/her problem. This would be a way to facilitate the patient's treatment adherence and in consequence improve the effectiveness of the AD treatment. In the present study the differential efficacy of two ways of applied homework assignments for the treatment of AD is explored with a between subject randomized controlled trial. After the evaluation phase, all participants receive a 6-8 sessions weekly CBT program. After each treatment session, they practice their assigned homework (using TEO or in the Traditional way) and they assess several clinical variables. After treatment completion, a post-treatment assessment will be carried out as well as follow-up assessments at 6- and 12-month.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* To meet current DSM-IV-TR criteria for Adjustment Disorder
* Be able to use a computer and having an Internet connection at home.

Exclusion Criteria:

* A severe mental disorder on Axis I: abuse or dependence of alcohol or other substances, psychotic disorder or Schizophrenia.
* A severe personality disorder or illness
* Presence of risk suicide
* Be receiving other psychological treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Beck Depression Inventory II (BDI-II) (Beck, Steer, & Brown, 1996) | 12 months
  BDI-II is one of the most widely used questionnaires to evaluate the severity of depression in pharmacological and psychotherapy trials. It consists of 21 items about the different symptoms characterizing the major depression disorder, summed to obtain the total score, which can be a maximum of 63 points. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and a test-retest reliability of around 0.8.
Change in Self-efficacy before and after homework assignment (Labpsitec 2010) | 2 months
  The participant assesses perceived self-efficacy to cope with her problem before and after practicing the homework assigned in both conditions (TEO and Traditional) in a scale from 1= "Nothing at all" to 7= "Totally".
Change in Inventory of Stress and Loss (Mor, Molés, Rachyla and Quero, 2015) | 12 months
  It is an adaptation of the Complicated Grief Inventory (CGI; Prigerson, 1995). It includes 17 items that assess to which extent the lost person/situation interferes in the individual's life on a scale ranging from 0 ("Never") to 4 ("Always"). The instrument has excellent internal consistency (Cronbach's alpha 0.86) and a test-retest reliability of around 0.9.

SECONDARY OUTCOMES:
Change in Posttraumatic Growth Inventory (PTGI) (Tedeschi y Calhoun, 1996) | 12 months
  - It is an instrument that assesses positive outcomes reported by people who have experienced a traumatic event. For each of the statements, participants indicate the degree to which this change occurred in their life as a result of their crisis, using the scale ranging from "I did not experience this change as a result of my crisis" (scored 0), to ''I experienced this change to a very great degree as a result of my crisis" (scored 5). The instrument has an excellent internal consistency (Cronbach's alpha 0,90) and acceptable test-retest reliability of around 0.71.
Change in Avoidance, Emotional Distress and Belief Scales (Adapted from Marks and Mathews 1979). | 12 months
  This instrument establishes the main situations and behaviors evoking distress, the intrusive thoughts or images, the predominant negative emotions, and the irrational thoughts related to the stressor event. The patient assesses using 0-10 scales (0= "Nothing at all"; 10= "Totally") the degree of avoidance and distress related to the situations/behaviors, thoughts/images, and emotions, as well as the degree of belief in the irrational thoughts
Change in Mood State before and after homework assignments (Labpsitec 2010) | 2 months
  The participant assesses mood state before and after practicing the homework assigned in both conditions (TEO and Traditional) on a 7-point Likert scale using faces reflecting different mood states.

OTHER OUTCOMES:
Change in Positive and Negative Affect Scale (PANAS) (Sandín et al., 1999). | 12 months
  The PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is from 10 to 50. The Spanish version has demonstrated high internal consistency (0.89 to 0.91 for PA and NA, respectively, in women, and 0.87 and 0.89 for PA and NA, respectively, in men) in college students (Sandín et al., 1999)
Change in Interference /Severity Scale rated by the Therapist (Adapted from ADIS-IV Interview by Di Nardo, Brown and Barlow 1994). | 12 months
  The therapist makes a global evaluation of the patient's interference and severity on a scale from 0 ("No impaired or without symptoms") to 8 ("Severely impaired or Very severe").

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Quero, Lecturer, Study Director — University Jaume I, Castellón, Spain; Maria del Mar Molés, Phd Student, Study Chair — University Jaume I, Castellón, Spain
Locations (1):
- University Jaume I, Catellon, Castellon, Spain

REFERENCES:
- [Background] Quero S, Botella C, Andreu-Mateu S, Baños R, Molés M. An adaptative Virtual Reality System for the treatment of Adjustment Disorder: 12-Months follow-up efficacy (November 2013). Symposium presented in ABCT's 47th Annual Convention. Nashville (EE.UU).
- [Background] Rochlen AB, Zack JS, Speyer C. Online therapy: review of relevant definitions, debates, and current empirical support. J Clin Psychol. 2004 Mar;60(3):269-83. doi: 10.1002/jclp.10263. PMID 14981791
- [Background] Beck, J. y Tompkins, M. Handbook of Homework Assignments in Psychotherapy. Nueva York. Springer. 2007
- [Background] Botella C, Baños R.M & Guillén V. Creciendo en la adversidad. Una propuesta de tratamiento para los trastornos adaptativos. In C. Vázquez & G. Hervás (Eds.), Psicología Positiva aplicada. Bilbao: DDB, 2008.
- [Background] Quero S, Moles M, Perez-Ara MA, Botella C, Banos RM. An online emotional regulation system to deliver homework assignments for treating adjustment disorders. Stud Health Technol Inform. 2012;181:273-7. PMID 22954870
- [Background] Baños, R. M., Guillen, V., Quero, S., García-Palacios, A., Alcaniz, M., & Botella, C. (2011). A virtual reality system for the treatment of stress-related disorders: A preliminary analysis of efficacy compared to a standard cognitive behavioral program. International Journal of Human-Computer Studies, 69 (9) 602-613.
- [Background] Quero, S., Andreu-Mateu, S., Moragrega, I., Baños, R.M., Molés, M., Nebot, S. y Botella, C. (en revisión). Un Programa Cognitivo-Conductual que utiliza la Realidad Virtual para el Tratamiento de los Trastornos Adaptativos: Una Serie de casos. Revista Argentina de Psicología Clínica (en prensa)
- [Background] Andreu-Mateu, S., Botella, C., Quero, S., Guillen, V., & Baños, R. (2012). La utilización de la realidad virtual y estrategias de psicología positiva en el tratamiento de los trastornos adaptativos. Behavioral Psychology/ Psicologia Conductual, 20 (2) 323-348.
- [Background] Casey P. Adjustment disorder: new developments. Curr Psychiatry Rep. 2014 Jun;16(6):451. doi: 10.1007/s11920-014-0451-2. PMID 24748555
- [Background] Maercker A, Brewin CR, Bryant RA, Cloitre M, van Ommeren M, Jones LM, Humayan A, Kagee A, Llosa AE, Rousseau C, Somasundaram DJ, Souza R, Suzuki Y, Weissbecker I, Wessely SC, First MB, Reed GM. Diagnosis and classification of disorders specifically associated with stress: proposals for ICD-11. World Psychiatry. 2013 Oct;12(3):198-206. doi: 10.1002/wps.20057. PMID 24096776
- See also: Laboratory of Psychology and Technology of the University Jaume I — http://www.labpsitec.uji.es
- See also: American Psychological Association — http://www.apa.org